CLINICAL TRIAL: NCT06585891
Title: VRC 617: A Phase 1, Open-Label, Dose-Escalation Study to Evaluate Safety and Pharmacokinetics of a Human Bispecific Antibody, VRC-HIVMAB0121-00-AB (CAP256J3LS) Administered Intravenously or Subcutaneously to Healthy Adults
Brief Title: Study of a Human Bispecific Antibody VRC-HIVMAB0121-00-AB (CAP256J3LS) Administered Intravenously or Subcutaneously to Healthy Adults
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 10001965; 001965-I
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01-15

CONDITIONS: HIV Infection
Keywords: Immune Response; HIV; Bi-Specific Antibody
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1 (Experimental): 5 mg/kg IV- single administration
  Interventions: Biological: VRC-HIVMAB0121-00-AB
- Group 2 (Experimental): 5 mg/kg SC- single administration
  Interventions: Biological: VRC-HIVMAB0121-00-AB
- Group 3 (Experimental): 20 mg/kg IV- single administration
  Interventions: Biological: VRC-HIVMAB0121-00-AB
- Group 4 (Experimental): 40 mg/kg IV- single administration
  Interventions: Biological: VRC-HIVMAB0121-00-AB
- Group 5 (Experimental): 5 mg/kg SC- repeat dosing
  Interventions: Biological: VRC-HIVMAB0121-00-AB
- Group 6 (Experimental): 20 mg/kg IV-repeat dosing
  Interventions: Biological: VRC-HIVMAB0121-00-AB

INTERVENTIONS:
Biological: VRC-HIVMAB0121-00-AB — The CAP256J3LS bispecific antibody (bsAbs) targets the V2-apex and CD4-binding sites of the HIV-1 envelope. It is composed of the light chain of CAP256V2LS, linked to the llama nanobody J3, which has broad CD4-binding site-directed neutralization.

SUMMARY:
Background:

HIV (human immunodeficiency virus) is the virus that causes AIDS (acquired immunodeficiency syndrome). Researchers want to find new ways to treat or prevent HIV infection. CAP256J3LS is a new product that uses antibodies. Antibodies are naturally occurring proteins; they target and disable disease-causing agents such as viruses. This new product may be able to stop HIV infections.

Objective:

To test the safety of CAP256J3LS in healthy people.

Eligibility:

People aged 18 to 60 years in good general health.

Design:

CAP256J3LS can be administered in 2 ways: (1) by a shot under the skin into the belly fat or (2) through a tube inserted into a vein in the arm. Participants will be divided into 6 groups: The study will open with the lowest dose of study product. The dose groups are spaced out to allow the study team to look over the safety data in each group. If there are no safety concerns in the lowest dose, then the next higher dose groups will be enrolled. This pattern will continue until all dose groups are enrolled.. Also, some participants will receive only 1 dose; others will receive 3 doses, each spaced 12 weeks apart.

Those who receive only 1 dose of the study drug will have 14 clinic visits over 6 months. Those who get 3 doses will have 27 visits over 11 months. Participants will provide blood samples at each visit. Urine samples may also be needed.

All participants will get a thermometer and a measuring tool. They will measure any redness, swelling, or bruising they have at the injection site. They will check their temperature every day for 7 days after receiving the study drug. They will record their highest temperatures and any symptoms they have.

...

DETAILED DESCRIPTION:
Design:

This first-in-human, Phase 1, open-label study will examine safety, tolerability, dose, and pharmacokinetics (PK) of CAP256J3LS (VRC-HIVMAB0121-00-AB) in healthy adults in a dose-escalation design. The primary hypothesis is that subcutaneous (SC) and intravenous (IV) administrations of CAP256J3LS will be safe and well-tolerated in healthy adults. A secondary hypothesis is that CAP256J3LS will be detectable in human sera with a definable half-life.

Study Products:

The CAP256J3LS bispecific antibody (bsAb) targets the V2-apex and CD4-binding sites of the HIV-1 envelope. It is composed of the J3 camelid nanobody linked to CAP256V2LS through a 15 amino acid linker arm attached to the N-terminus of the CAP256V2LS light chain. The addition of the J3 nanobody adds a CD4-binding site directed neutralization functionality to the CAP256V2LS, which targets the V2 region of the HIV Env trimer. The bispecific antibody was developed by the VRC/NIAID/NIH and is manufactured under cGMP regulations at the VRC Pilot Plant operated under contract by the Vaccine Clinical Materials Program (VCMP), Leidos Biomedical Research, Inc., Frederick. MD.

Participants:

Healthy adults, 18-60 years of age

Study Plan:

This open-label study will include 6 groups to evaluate CAP256J3LS administered one time or by repeat dosing. Enrollment will begin with the 5 mg/kg dose groups, and enrollment for subsequent dose groups will proceed after dose-escalation safety reviews. Assessment of safety will include solicited reactogenicity and other adverse events, clinical observations, and monitoring of hematological and chemistry parameters at clinical visits throughout the study.

ELIGIBILITY:
* INCLUSION CRITERIA:

A participant must meet all of the following criteria:

1. Willing and able to complete the informed consent process.
2. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
3. Available for clinical follow-up through the last study visit.
4. 18 to 60 years of age.
5. In good general health without a clinically significant medical history.
6. Physical examination without clinically significant findings within the 56 days prior to enrollment.
7. Adequate venous access if assigned to an IV group or adequate abdominal subcutaneous tissue if assigned to a SC group.
8. Willing to have blood samples collected, stored indefinitely, and used for research purposes.

   Laboratory Criteria within 56 days prior to enrollment:
9. White blood cell count (WBC): 2,500-12,000/mm^3.
10. WBC differential either within institutional normal range or accompanied by the Principal Investigator (PI) or designee approval, excluding absolute lymphocyte count which must not be lower than normal range.
11. Platelets: 125,000 - 400,000/mm^3.
12. Hemoglobin within institutional normal range or is lower than normal range but does not meet Grade 1 criteria and is not clinically concerning.
13. Creatinine: <= 1.1 x Upper Limit of Normal (ULN).
14. ALT: <= ULN.
15. AST: <= ULN.
16. ALP: <= ULN.
17. Total bilirubin within institutional normal range or is outside normal range but does not meet Grade 1 criteria and is not clinically concerning
18. Direct bilirubin: <= ULN
19. Negative HIV 1/2 Antibody/Ag test.

    Female-Specific Criteria:
20. Agrees to use an effective means of birth control from 21 days prior to enrollment through the duration of study participation.
21. Negative beta-HCG (human chorionic gonadotropin) pregnancy test (urine or serum) on day of enrollment for women presumed to be of reproductive potential.

EXCLUSION CRITERIA:

A participant will be excluded if one or more of the following conditions apply:

1. Woman who is breast-feeding or planning to become pregnant during study participation.
2. Weight > 115 kg.
3. Any history of a severe allergic reaction with generalized urticaria, angioedema or anaphylaxis prior to enrollment that has a reasonable risk of recurrence during the study.
4. Hypertension that is not well controlled.
5. Receipt of any investigational study product within 28 days prior to enrollment.
6. Receipt of an investigational HIV vaccine or anti-HIV monoclonal antibody.
7. Receipt of any live attenuated vaccine within 28 days prior to enrollment.
8. Receipt of any vaccine within 2 weeks prior to enrollment.
9. Known history of Gilbert's syndrome.
10. Known history of kidney or liver disease.
11. Diabetes mellitus (type I or II), with the exception of a history of gestational diabetes.
12. More than 10 days of systemic immunosuppressive medications or cytotoxic medications within the 4 weeks prior to enrollment or any within 14 days prior to enrollment.
13. Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.
14. Any other chronic or clinically significant medical condition that in the opinion of the investigator would jeopardize the safety or rights of the volunteer, including but not limited to diabetes mellitus, hepatitis, asthma, infectious disease, autoimmune disease, psychiatric disorder, heart disease, cancer and clinically significant forms of drug or alcohol abuse.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2026-06-09 (Estimated); Study Completion 2027-06-09 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of CAP256J3LS (5 mg/kg SC) administered to healthy adults | Through 24 weeks after product administration
  To evaluate the safety and tolerability of a single SC dose
Safety and tolerability of CAP256J3LS ( 5mg/kg or 20mg/kg or 40 mg/kg IV) administered to healthy adults | Through 24 weeks after product administration
  To evaluate the safety and tolerability of a single IV dose
Safety and tolerability of CAP256J3LS ( 5 mg/kg SC) administered for for a total of 3 injections in 12 week intervals to healthy adults | Through 24 weeks after last product administration
  To evaluate the safety and tolerability of a repeat SC dosing
Safety and tolerability of CAP256J3LS ( 20 mg/kg IV) administered for for a total of 3 injections in 12 week intervals to healthy adults | Through 24 weeks after last product administration
  To evaluate the safety and tolerability of a repeat IV dosing

SECONDARY OUTCOMES:
PK will be evaluated at each dose level and route of administration | Throughout the study
  To evaluate the pharmacokinetics of CAP256J3LS

CONTACTS AND LOCATIONS:
Overall Officials: Lasonji A Holman, C.R.N.P., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang B, Gorman J, Kwon YD, Pegu A, Chao CW, Liu T, Asokan M, Bender MF, Bylund T, Damron L, Gollapudi D, Lei P, Li Y, Liu C, Louder MK, McKee K, Olia AS, Rawi R, Schon A, Wang S, Yang ES, Yang Y, Carlton K, Doria-Rose NA, Shapiro L, Seaman MS, Mascola JR, Kwong PD. Bispecific antibody CAP256.J3LS targets V2-apex and CD4-binding sites with high breadth and potency. MAbs. 2023 Jan-Dec;15(1):2165390. doi: 10.1080/19420862.2023.2165390. PMID 36729903
- [Background] McCoy LE, Quigley AF, Strokappe NM, Bulmer-Thomas B, Seaman MS, Mortier D, Rutten L, Chander N, Edwards CJ, Ketteler R, Davis D, Verrips T, Weiss RA. Potent and broad neutralization of HIV-1 by a llama antibody elicited by immunization. J Exp Med. 2012 Jun 4;209(6):1091-103. doi: 10.1084/jem.20112655. Epub 2012 May 28. PMID 22641382
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001965-I.html